

# TRIAL STATISTICAL ANALYSIS PLAN

(Part 1 of 1368-0098)

| <b>Document No.:</b> | c4342178 | 87-01 |
|---|---|---|
| BI Trial No.: | 1368-0098 | |
| Title: | Randomised, double-blind, placebo-controlled, study to evaluate the efficacy and safety of spess with moderate to severe hidradenitis suppuratival | olimab in patients |
| Investigational Product(s): | Spevigo®, spesolimab | |
| Responsible trial statistician(s): | Tel.: Fax: | |
| Date of statistical analysis plan: | 13-08-2024 | |
| Version: | 1.0 | |
| | Proprietary confidential information eim International GmbH or one or more of its affiliated compani full or in part - be passed on, reproduced, published or otherwise used without | |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 1. TABLE OF CONTENTS

| TITLE | PAGE | 1 |
|---|---|---|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 9 |
| 5.<br>5.1<br>5.2<br>5.2.1<br>5.2.2 | ENDPOINT(S) | 11<br>11 |
| 6. | GENERAL ANALYSIS DEFINITIONS | 17 |
| 6.1 | TREATMENT(S) | 17 |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | INTERCURRENT EVENTS | |
| 6.4 | SUBJECT SETS ANALYSED | 20 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 23 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 28 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTIC | CS28 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 29 |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY OBJECTIVE ANALYSIS | 30 |
| 7.4.1 | Main analysis | 30 |
| 7.5 | SECONDARY OBJECTIVE ANALYSIS | 35 |
| 7.5.1 | Key secondary objective analysis | 35 |
| 7.5.2 | Secondary objective analysis | |

c43421787-01

| Pror | rietary | confidential | Informatio | n © 2024 | Roehringer | Ingelheim | International | GmbH or one | e or more of its | affiliated | companies |
|---|---|---|---|---|---|---|---|---|---|---|---|

| • | | • |
|--------------|-----------------------------------------------|----|
| 7.7 | EXTENT OF EXPOSURE | 38 |
| <b>7.8</b> | SAFETY ANALYSIS | 38 |
| 7.8.1 | Adverse Events | 38 |
| 7.8.2 | Laboratory data | 41 |
| 7.8.3 | Vital signs | 44 |
| 7.8.4 | ECG | 44 |
| 7.8.5 | Local Tolerability | 44 |
| 7.8.6 | Acne Episodes | |
| <b>7.9</b> | OTHER ANALYSIS | 45 |
| <b>7.9.1</b> | Biomarker analyses | 45 |
| <b>7.9.2</b> | PK / PD analyses | 45 |
| 7.9.3 | Immunogenicity | 46 |
| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION | 47 |
| 9. | REFERENCES | 48 |
| 11 | HISTORY TARLE | 64 |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## LIST OF TABLES

Date: 07-08-2024, Version 1.0

| Table 6.1: 1 | Flow chart of analysis periods of the study according to randomized | |
|---|---|---|
| | treatment (Part 1 – Phase IIb) | 17 |
| Table 6.3: 1 | Summary of intercurrent events and handling strategy for primary endpoint. | 19 |
| Table 6.3: 2 | Summary of intercurrent events and handling strategy for continuous | |
| | secondary and further endpoints | 19 |
| Table 6.3: 3 | Summary of intercurrent events and handling strategy for binary further | |
| | endpoints and time-to-event endpoints | 20 |
| Table 6.4: 1 | Subject sets analyzed | 22 |

| Table 7.1: 1 | Categories for demographic variables and baseline characteristics | 29 |
|---|---|---|
| Table 7.4: 1 | Total dose per treatment arm | 32 |
| | Contrast coefficients | |
| Table 7.8.1: 1 | Project MEDDRA search criteria for User Defined Adverse Events | |
| | Concepts | 40 |
| Table 11: 1 | History table | 64 |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 2. LIST OF ABBREVIATIONS


| Term | Definition / description |
|---|---|
| ADA | Anti-drug antibodies |
| ADS | Analysis dataset |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALQ | Above the upper limit of quantification |
| ALT | Alanine aminotransferase |
| AdT | Abscess and draining tunnel |
| AN | Abscess and inflammatory nodule |
| ANdT | Abscess, inflammatory nodule and draining tunnel |
| AP | Alkaline phosphatase |
| AST | Aspartate aminotransferase |
| ATC3 | Anatomical-Therapeutic-Chemical classification level 3 |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BMI | Body mass index |
| BSA | Body surface area |
| CARE | Clinical data analysis and reporting environment |
| CGI | Clinical Global Impression |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CRF | Case report form |
| CRP | C-reactive protein |
| CTIS | Clinical Trials Information System |
| CTP | Clinical trial protocol |
| CTR | Clinical trial report |
| CV | Arithmetic coefficient of variation |
| DBLM | Database lock meeting |
| DNA | Deoxyribonucleic acid |

c43421787-01

| Term | Definition / description |
|---|---|
| dT | Draining fistula/tunnel |
| EC | Estimand concept |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EMA | European Medicines Agency |
| ES | Enrolled set |
| FACIT | Functional Assessment of Chronic Illness Therapy |
| FUP | Follow-up |
| gCV | Geometric coefficient of variation |
| GCP | Good Clinical Practice |
| gMean | Geometric mean |
| GPP | Generalized pustular psoriasis |
| HASI | HS Area and Severity Index |
| HS | Hidradenitis suppurativa |
| HS-PGA | HS Physician Global Assessment |
| HiSCR | Hidradenitis suppurativa clinical response |
| mHiSCR | Modified - Hidradenitis suppurativa clinical response |
| HS-CRP | High-Sensitivity C-Reactive Protein |
| IHS4 | International Hidradenitis Suppurativa Severity Score System |
| IL-36 | Interleukin 36 |
| IL-36R | Interleukin 36 Receptor |
| NRS | numerical rating scale |
| ICH | International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use |
| HiS-QoL | Hidradenitis suppurativa quality of life |
| iPD | Important protocol deviation |
| ICEs | Intercurrent events |
| i.v. | intravenous |
| MedDRA | Medical Dictionary for Regulatory Activities |
| DLQI | Dermatology Life Quality Index |
| NRI | No response imputation |
| OC | Observed cases |

c43421787-01

| Term | Definition / description |
|-------|----------------------------------------|
| OR | Original results |
| OLE | Open Label Extension |
| PD | Pharmacodynamic(s), protocol deviation |
| PE | Primary endpoint |
| PK | Pharmacokinetic(s) |
| PKS | Pharmacokinetic parameter set |
| PPS | Per protocol set |
| PT | Preferred term |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| RAGe | Report appendix generator |
| REP | Residual effect period |
| RNA | Ribonucleic acid |
| RPM | Report planning meeting |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SDL | Subject data listing |
| SI | Système international d'unités |
| SOC | System organ class |
| TS | Treated set |
| TSAP | Trial statistical analysis plan |
| UDAEC | User-defined Adverse Event Category |
| ULN | Upper limit of normal range |
| VAS | Visual analogue scale |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 3. INTRODUCTION

This TSAP describes the statistical analyses for Part 1 of study 1368-0098.

As per ICH E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization. In this TSAP, subject and patient will be used interchangeably.

SAS® Version 9.4 will be used for all analyses.

## For Part 1 (Phase IIb):


Per CTP, the primary and interim analysis for Part 1 will be conducted after the last trial participant completes the Week 8 visit and Week 16 visit respectively. Separate iDBLs will be performed for primary and interim analysis and a respective team ("shadow team") independent of the main trial team will be formed to conduct the necessary analyses and ensure to maintain the blind and restrict access to the randomization codes from the main trial team for both primary and interim analysis. Details of this process will be described in a separate data logistics plan which will also specify details on data access.

Analyses of the skin and blood biomarkers will be described in a separate biomarker SAP, unless otherwise specified in this document.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses stated in the CTP (latest version) will be performed as planned with the following adaptations.

The below further efficacy endpoints have been updated:

- Achievement of HiSCR50 at each scheduled assessment.
   HiSCR50 is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase in the abscess or draining fistula count.
- Absolute change from baseline in Patient Global Impression of Change (PGI-C) score over time.

This endpoint will be updated to:

Patient Global Impression of Change (PGI-C) score at each scheduled assessment over time.

• Absolute change from baseline in Patient Global Impression of Severity (PGI-S) score over time.

This endpoint will be updated to:


Patient Global Impression of Severity (PGI-S) score at each scheduled assessment over time.

The below further efficacy endpoints, which were not specified in the CTP version 2.0, have been added:

- Achievement of HiSCR75 at each scheduled assessment.
   HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase in the abscess or draining fistula count.
- Achievement of HiSCR90 at each scheduled assessment.
   HiSCR90 is defined as at least a 90% reduction from baseline in the total abscess and inflammatory nodule count, with no increase in the abscess or draining fistula count.
- Achievement of mHiSCR at each scheduled assessment: mHiSCR is defined as at least a 50% reduction in total ANdT count relative to baseline. and at least 50% reduction in total dT count relative to baseline.
- Achievement of mHiSCR-AdT at each scheduled assessment: mHiSCR-AdT is defined as at least a 50% reduction in the total AdT count with no increase in inflammatory nodule count, no increase in abscess count, and no increase in dT count relative to baseline.
- Achievement of mHiSCR-AdT(2) at each scheduled assessment: mHiSCR-AdT (2) is defined as at least 50% reduction in the total ANdT count relative to baseline and at least 50% reduction in total AdT count relative to baseline.

## Boehringer Ingelheim TRIAL STATISTICAL ANALYSIS PLAN 1368-0098


c43421787-01

- Achievement of 2 points reduction in Physician's Global Assessment (PGA) score from baseline at each scheduled assessment (only for patients with a PGA  $\geq$  2 at baseline).
- Achievement of at least 30% reduction from Week 1 measurement in Numerical rating scale in Patient's Global Assessment of HS pain at each scheduled assessment.
- Percent change from baseline in Numerical rating scale in Patient's Global Assessment of HS pain at each scheduled assessment
- Percent change from Week 1 in Numerical rating scale in Patient's Global Assessment of HS pain at each scheduled assessment

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 5. ENDPOINT(S)

## **5.1 PRIMARY ENDPOINT(S)**

The primary endpoint of the study is defined in CTP as:

Part 1 (Phase IIb): Percent change from baseline in dT count at Week 8

## **5.2 SECONDARY ENDPOINT(S)**

#### 5.2.1 Key secondary endpoint(s)

Part 1 (Phase IIb): Not applicable

## 5.2.2 Secondary endpoint(s)

## Part 1 (Phase IIb) Efficacy


- Percent change from baseline in dT count at Week 16.
- Absolute change from baseline in IHS4 value at Week 8.
- Absolute change from baseline in IHS4 value at Week 16.

## Safety

Occurrence of treatment emergent adverse events (TEAEs)



c43421787-01



c43421787-01



c43421787-01



c43421787-01



c43421787-01



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 6. GENERAL ANALYSIS DEFINITIONS

## **6.1 TREATMENT(S)**

## Part 1 (Phase IIb)


The analysis periods are defined relative to the day of randomization (Day 1) in <u>Table 6.1:1</u>:

Table 6.1: 1 Flow chart of analysis periods of the study according to randomized treatment

| Study analysis period | Description | Start (included) | End (included) |
|---|---|---|---|
| Screening period | Screening | Earliest of (Date of informed consent, first screening procedure) | Date/time of start of the first study dose minus 1 minute. |
| Loading period<br>(from Day 1 to | On-<br>treatment<br>period | Date/time of start of<br>the first study<br>loading dose (Day<br>1) | Earliest of i) Date/time of start of the first maintenance dose minus1 minute; ii) Date of end of last loading dose + 112 days at 11:59 p.m. if patient early discontinued study treatment before visit; iii) last contact date on End of Study page at 11:59 p.m. |
| Maintenance<br>period I (from<br>to<br>Week 8) | | Date/time of start of<br>the first<br>maintenance dose<br>for visit (if<br>applicable) | Earliest of i) Date/time of start of the study maintenance dose for Week 8 visit minus 1minute; ii) Date of end of last maintenance dose + 112 days at 11:59 p.m. if patient early discontinued study treatment before Week 8 visit; iii) last contact date on End of Study page at 11:59 p.m. |
| Maintenance<br>period II (from<br>Week 8 to<br>Week 16) | | Date/time of start of<br>the study<br>maintenance dose<br>for Week 8 visit (if<br>applicable) | Earliest of i) Date/time of start of the study maintenance dose for Week 16 visit minus 1minute; ii) Date of end of last maintenance dose + 112 days at 11:59 p.m. if patient early discontinued study treatment before Week 16 visit; iii) last contact date on End of Study page at 11:59 p.m. |
| Maintenance<br>period III (from<br>Week 16 to | | Date/time of start of<br>the study<br>maintenance dose<br>for Week 16 visit (if<br>applicable) | Earliest of i) Date/time of the first treatment in OLE trial 1368.0130 minus1 minute if subject is rolled over; ii) Date of end of last maintenance dose + 112 days at 11:59 p.m. if patient early discontinued study treatment; iii) last contact date on End of Study page at 11:59 p.m. |
| Off-treatment<br>phase <sup>1</sup> (if<br>applicable) | Off-<br>treatment<br>period | Date of end of last<br>study dose + 113<br>days at 0:00 a.m. | Latest of i) Date of EOS visit; ii) last contact date on End of Study page at 11:59 p.m. |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Dates are defined individually per patient. If more than one date is associated with a specific visit, measurements associated with a specific date are assigned to a study analysis period according to the rules specified in the table. An analysis period will not extend beyond the start date of the following phase. 

<sup>1</sup> The off-treatment period only exists for patients who early discontinued study treatment or choose not to enter the extension study 1368-0130, whose last contact date is after the date of end of last study treatment + 112 days.

The following labels for the treatment groups for all analysis is according to the randomized treatment up to Visit 14 (Week 16):

| • | receive placebo); |
|---|-------------------|
| • | "Speso Low" ( |
| | [Week 16]); |
| • | "Speso Medium" |
| | [Week 16]); |
| • | |
| | [Week 16]): |

- "Speso Total" (i.e. randomised to any of the spesolimab group);
- "Overall Total" (i.e. randomised to any treatment group regardless of placebo or Spesolimab group).

#### **6.2 IMPORTANT PROTOCOL DEVIATIONS**

Each protocol deviation must be assessed to determine whether it is an important protocol deviation(iPD). For definition of iPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (iPD)" (9.6).

Handling of iPDs in analysis is included in the DV domain specifications and stored within the Trial Master File (TMF) in Electronic Document Management System (EDMS). iPDs may lead exclusion of subjects from the Per-Protocol set (PPS), which will be specified in DV domain specifications.

#### 6.3 INTERCURRENT EVENTS

The expected intercurrent events of interest in this trial are:

Use of rescue medication

Treatment discontinuation due to AE/lack of efficacy

Treatment discontinuation due to other reasons, e.g. relocating or other logistical reasons.

Use of restricted medication

Death


The strategies for handling intercurrent events up to Week 16 visit are as follows:

- Treatment policy (ET): Use of "treatment policy" approach disregards the intercurrent event and uses the value of the variable regardless of the occurrence of the intercurrent event.
- Hypothetical approach (EH): Data after the intercurrent events will be censored.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

- Composite strategy (EC): Use of composite approach, where data after the intercurrent events were treated as a non-responder.

If multiple intercurrent events occur to the same patient up to Week 16 visit, the intercurrent event with composite strategy will be considered.

Summary of intercurrent events and handling strategy for primary endpoint are listed in <u>Table 6.3: 1</u>.

Table 6.3: 1 Summary of intercurrent events and handling strategy for primary endpoint

| Intercurrent Events | Primary Estimand (ET) | Supplementary Estimand (EH) |
|---|---|---|
| Use of rescue medication | ET | EH (Censor*) |
| Treatment discontinuation due to AE/lack of efficacy | ET | EH (Censor*) |
| Treatment discontinuation due to other reasons | ET | EH (Censor*) |
| Use of restricted medication | ET | EH (Censor*) |
| Death | ЕН | EH (Censor*) |

<sup>\*</sup>Data after the time when intercurrent event happens will be censored.


Summary of intercurrent events and handling strategy for **continuous secondary and further endpoints** are listed in Table 6.3: 2.

Table 6.3: 2 Summary of intercurrent events and handling strategy for continuous secondary and further endpoints

| Intercurrent events | Primary Estimand (ET) |
|------------------------------------------------------|-----------------------|
| Use of rescue medication | ET |
| Treatment discontinuation due to AE/lack of efficacy | ET |
| Treatment discontinuation due to other reasons | ET |
| Use of restricted medication | ET |
| Death | EH |

1368-0098

c43421787-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Summary of intercurrent events and handling strategy for **binary further endpoints** are listed in Table 6.3: 3.

Table 6.3: 3 Summary of intercurrent events and handling strategy for binary further endpoints

| Intercurrent events | Primary Estimand (EC-ET) |
|---|---|
| Use of rescue medication | EC |
| Treatment discontinuation due to AE/lack of efficacy | ET |
| Treatment discontinuation due to other reasons | ET |
| Use of restricted medication | EC |
| Death | EC |

Primary Imputation Approach for binary endpoints – No Response Imputation [NRI]:

- If there are data at visits both before and after the visit with a missing outcome, then impute as success only if both neighbouring visits also represent a success (independent of whether the preceding and following observations were selected for analysis based on time windows described in <a href="Section 6.7">Section 6.7</a> and no rescue treatment has been given during this period).
- Otherwise, impute as a failure.

## 6.4 SUBJECT SETS ANALYSED

The following analysis sets will be defined for statistical analyses:

## Enrolled Set (ES):

This patient set includes all patients who signed informed consent. The ES will be used for the analyses of patient disposition.

#### Randomized Set (RS):

This patient set includes all patients who were randomized in the trial. Treatment assignment will be as randomised. It will be used for analyses of subject for baseline demographics, disease characteristics and iPD etc.

#### Full Analysis Set (FAS):


This patient set includes all randomized patients and received at least one dose of study drug. This is the main analysis set for presentation of efficacy data. Patients will be analysed according to their planned treatment group.

#### • Full Analysis Set (FAS-Post16):

This patient set includes all randomized patients and received at least one dose of study drug during the maintenance period III (from Week 16 to set for presentation of efficacy data post week 16.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### Safety Analysis Set (SAF):

1368-0098

This subject set includes all subjects who were randomized and received at least one dose of study drug. This is the main analysis set for safety. Subjects will be analysed according to the actual treatment received at Day 1.

#### Per-Protocol Set (PPS):

This subject set includes all subjects in the randomized set who adhered to the CTP without any iPDs which are flagged for exclusion from the PPS. The PPS will be used for sensitivity analysis on the primary endpoint.

The discussion of all exceptional cases and problems and the decisions on the allocation of patients to populations will be made at latest at the DBLM. A separate DBLM will be performed prior to each database snapshot of this trial.

### PK Parameter Analysis Set (PKS) (if applicable):

This patient set includes all patients in the RS who provide at least one evaluable observation for the Spesolimab concentration, which was not flagged for exclusion. The PKS will be used for the display of concentrations.

#### ADA Analysis Set:


This patient set includes all patients in the RS who provide baseline and at least one reportable post-baseline ADA data.

#### Biomarker Set (BMS) (if applicable):

This patient set includes all patients in the RS who have analyzable data (observed or imputed) in at least one biomarker.

#### **Handling of Treatment Misallocations in Analysis Sets**

If a subject is treated but not randomized, they will be excluded from the efficacy analysis and safety analysis by definition. However, subjects under such circumstances will be described in the final clinical trial report.

If a subject is randomized but takes incorrect treatment during the study, then:

- For efficacy analyses according to RS and PPS, they will be reported under their randomized treatment groups.
  - O In the case of stratification error at randomization, the subjects will be analyzed according to the stratum to which they actually belong to (regardless of any mis-assignment to treatment based on identification of the wrong stratum from IRT), as such an error occurs before randomization and is therefore consistent with regulatory guidance.
- For the safety analysis based on SAF, the actual treatment will be used as below:

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

- o If a subject is planned to receive administration of Spesolimab (randomized to Speso) at day 1, then patients will be reported under their randomized treatment group for safety analysis because the overall safety profile is expected to be driven by the amount of Spesolimab received in totality over the entire treatment duration. It is not expected that the safety profile will deviate from the planned treatment regimen if the subject receives only a few vials of the incorrect medication at only some dosing occasions.
- o If a subject is planned to receive placebo treatment at day 1, then they will be reported under the placebo arm if they are treated and receive no vial of randomized Spesolimab. If the subject receives >= 1 vial of randomized Spesolimab before week 16, then the patient will be handled differently for efficacy analysis and safety analysis. It will keep as placebo for efficacy reporting. For safety, then the patients will be reported as their treated Spesolimab group.

Table 6.4: 1 Subject sets analyzed

| Subject Set | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Class of endpoint | ES | RS | FAS | SAF | PPS | PKS | ADA | BMS |
| Disposition | X | | | | | | | |
| Demographic and baseline characteristics | | | X | | | | | |
| Baseline condition / Medical history | | | X | | | | | |
| Compliance and Exposure | | | | X | | | | |
| Concomitant medication/therapy | | | X | | | | | |
| iPD | | X | | | | | | |
| Primary endpoint | | | Xª | | $X^b$ | | | |
| Secondary endpoints | | | X | | | | | |
| Further endpoints | | | Xc | | | | | |
| Safety endpoints | | | | X | | | | |
| Concentration (if applicable) | | | | | | X | | |
| Anti-drug antibody | | | | | | | X | |
| Biomarker (if applicable) | | | | | | | | X |

a Primary analysis; b Sensitivity analysis; c FAS including FAS-post 16.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Section 7.3 of the CTP describes the handling of missing data.


Missing or incomplete AE dates are imputed according to BI standards (9.1). Missing data and outliers of PK data are handled according to BI standards (9.2).

For incomplete information on the date of first diagnosis, time since first diagnosis will be calculated as follows:

- If the year of first diagnosis is unknown, time since first diagnosis will be set to missing.
- If day and month of the first diagnosis are unknown, time since first diagnosis will be calculated as if diagnosed on the 30<sup>th</sup> June of that year.

c43421787-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

• If only the day of the first diagnosis is unknown, time since first diagnosis will be calculated as if diagnosed on the 15<sup>th</sup> of that month.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Unless otherwise specified, measurements reported with date and time and taken prior to start of administration of trial treatment will be considered pre-treatment values; measurements reported with a date only (and no time) and taken on the day of first administration of trial treatment will also be considered pre-treatment values. These pre-treatment values will be assigned to visits according to the nominal visit number as recorded on the eCRF or as provided by the laboratory.

Patient reported output (PRO) measurements reported prior to/on the date of the drug administration will be taken as pre-treatment values, regardless the time of measurements taken if there exist.

Baseline, unless otherwise specified, is defined as the last measurement collected prior to the start of administration of the trial treatment.

Measurements taken after start of administration of trial treatment will be considered either on- or off-treatment values based on the definition in <u>Section 6.1</u>, and will be assigned to visits for statistical analysis, if applicable, as defined below.

Analysis of AE data, potentially clinically significant abnormal laboratory values, concomitant medication or non-drug therapies, as well as use of rescue medication will not be based on visits. Frequency tables for these data will be using on-treatment data and categorized based on their occurring/starting dates. Therefore, no assignment to time windows will be necessary for such data.

The derivation of the last value, minimum value and maximum value of laboratory and vital signs data will consider all on-treatment values (whether or not selected in any time window; see <u>Table 6.1: 1</u> for definition of the on-treatment period) within the period of interest; these will be derived for analysis of laboratory and vital signs data.

All other safety, efficacy and biomarker measurements will be assigned to visits based on extended time windows around the planned visit dates, defined relative to the day of first trial treatment (which is scheduled for Visit 2). These extended time windows are defined in <u>Table 6.7: 1</u> and <u>Table 6.7: 2</u>.

c43421787-01

c43421787-01



c43421787-01



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7. PLANNED ANALYSIS

The primary objective for dose finding Phase IIb (Part 1) are as follows:

- (1) to demonstrate a non-flat dose response curve, evaluate the quantitative treatment effect size, and evaluate the dose-response relationship based on the primary endpoint of percent change from baseline in dT count at Week 8;
- (2) to determine an optimal dose candidate for Part 2 by incorporating information of available safety and of efficacy based on the primary endpoint of percent change from baseline in dT count at Week 8.

The primary and interim analysis for Part 1 will be conducted after the last trial participant completes the Week 8 visit and Week 16 visit respectively. Final trial analysis is planned to be performed at the end of the study once all randomized patients have completed the study (including any follow-up period). If applicable, details of biomarker analyses will be provided in a separate Biomarker Statistical Analysis Plan.

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / SD / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to mean, standard deviation, minimum and maximum.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all subjects in the respective subject set regardless of whether they have non-missing values or not).

The precision for percentages should be one decimal point, unless the denominator is smaller than 100 (in all treatment columns), in which case percentages are given in integer numbers. The category missing will be displayed only if there are actually missing values.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.


Descriptive statistics will be presented by treatment for demographic variables and baseline characteristics, based on the FAS. More details could refer to Section 5.4.1.

For continuous demographic variables listed in <u>Table 7.1:1</u>, they will be presented by the number and percentage of patients in the categories defined in <u>Table 7.1:1</u>.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Table 7.1: 1 Categories for demographic variables and baseline characteristics

| · | |
|---|---|
| Variable | Categories |
| Age | < 30 years<br>30 to < 65 years<br>≥ 65 years |
| Weight | ≤60 kg<br>>60 to ≤90 kg<br>>90 kg |
| Weight based on popPK model # | <72kg<br>72 to ≤122kg<br>>122kg |
| BMI | < 25 kg/m2<br>25 to < 30 kg/m2<br>≥ 30 kg/m2 |
| Time since first diagnosis | <ul> <li>≤ 1 year</li> <li>&gt; 1 to ≤ 5 year</li> <li>&gt; 5 to ≤ 10 years</li> <li>&gt; 10 years</li> </ul> |
| Baseline dT count | |
| Neutrophil level | High > 7.23 X10^9 /L<br>Low ≤ 7.23 X10^9 /L |
| Baseline<br>neutrophil/lymphocyte<br>ratio | 1 to <=2 >2 to <=3 >3 |
| IHS4 severity | Mild: $\leq 3$<br>Moderate: $>3$ to $\leq 10$<br>Severe: $>10$ |

<sup>#</sup> The cut-off values of weight are based on the body weight values corresponding to the range of 80% to 125% of steady-state AUC0-  $\tau$  (any dosing regimen) using 94 kg as a reference, according to the population PK model.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION


Only descriptive statistics are planned for this section of the report.

Concomitant diseases (i.e., baseline conditions) and concomitant non-drug therapies will be coded according to the most recent version of Medical Dictionary for Drug Regulatory Activities (MedDRA). Concomitant medications will be coded according to the most recent version of the World Health Organization – Drug Dictionary (WHO-DD).

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Concomitant diseases which are present at start of the study will be descriptively summarized by treatment based on the FAS.

A medication/non-drug therapy will be considered concomitant to treatment, if it

- Is ongoing at the start of first study dose or
- Starts within the on-treatment period (see <u>Section 6.1</u> for the definition)

A medication/non-drug therapy will be considered as prior medication/non-drug therapy, if the end date of the medication/therapy is at any time prior to the start of first study dose.

Concomitant medication use (excluding rescue medication) taken at any time during the ontreatment period (cf. <u>Section 6.1</u>) will be summarized by treatment based on FAS, with frequency and percentage of patients by Anatomical Therapeutic Chemical 3 (ATC3) class and preferred name.

Concomitant use of non-drug therapies (excluding rescue therapy) taken any time during the on-treatment period (cf. <u>Section 6.1</u>) will be summarized by treatment based on FAS, with frequency and percentage of patients.

Use of rescue medication will be summarized separately based on FAS.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report. Treatment compliance (see <u>Section 5.4.2</u> for the definition and calculation) will be summarized by treatment and period on SAF using descriptive statistics (N, mean, SD, minimum, median, maximum).

#### 7.4 PRIMARY OBJECTIVE ANALYSIS

#### 7.4.1 Main analysis

#### Part 1 (Phase IIb)


The main analysis of the primary endpoint will use a treatment policy estimand. Details of handling the intercurrent events are addressed in Section 7.2.2 of the clinical trial protocol and Table 6.3.1. This main analysis of the primary efficacy endpoint will be performed on the full analysis set. Subjects will be analyzed according to the stratum to which they actually belong. Missing data will be handled using a mixed effects model with repeated measures (MMRM) under the assumption of missing at random.

The descriptions below are based on the primary objective and secondary objective, respectively.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### **Primary Objective: Dose Finding**

For the primary endpoint analysis, first a mixed effect model for repeated measurements (MMRM) is calculated to estimate the treatment effects and the corresponding covariance matrix. Using the MCPMod approach (9.4, 9.5), these estimates are then further used to

- (1) test for a non-flat dose response curve
- (2) identify suitable dose-response shapes out of a selection of candidate models.

The final dose-response model is derived as a weighted average over all significant model shapes. Planned total dose before Week 8 will be used to evaluate dose response curve.

Details on both the specification of the MMRM and the MCPMod approach are given in the CTP Section 7.2.2.

#### **MMRM** analysis

The % change in dT count from baseline (Visit 2), at Visits 4, 6, 8 and 10 ( , 8) will be evaluated using an MMRM accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, TNFi status at baseline and categorical baseline dT count at each visit. The unstructured covariance structure will be used to model the within patient measurements. To estimate denominator degrees of freedom the Kenward-Roger approximation will be used.

SAS code for MMRM for the endpoint of dT count:

PROC MIXED DATA=alldat cl method=reml;

CLASS dt\_base\_categorical visit trt TNFi subject;

MODEL ept = TNFi visit\*trt dt\_base\_categorical \*visit/ddfm=kr s CL;

REPEATED visit / subject= subject type=un r rcorr;

LSMEANS visit\*trt / pdiff=all om cl alpha=0.05 slice=visit;

RUN;

Results of the MMRM (N, mean, SE and 95% CI per dose group and timepoint) will be presented in tables and displayed graphically.

#### MCPMod Analysis


For the primary analysis the dose-response relationship will be modeled using the total doses. Here, the total is the sum of all doses administered to the patient prior to the week 8 visit including both loading and maintenance phase. Thereby, it is assumed that the cumulative concentrations over time (AUC) and thus the cumulative total dose is the key driver of the efficacy response in the modelling part of MCPMod. <u>Table 7.4: 1</u> shows the calculated total doses per treatment arm.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Table 7.4: 1 Total dose per treatment arm

| Treatment arm | Total dose |
|-----------------------------|-----------------------------|
| High dose regimen (Arm 1) | |
| | Total dose: Spesolimab |
| Medium dose regimen (Arm 2) | |
| | Total dose: Spesolimab |
| Low dose regimen (Arm 3) | |
| | Total dose: Spesolimab |
| Placebo (Arm 4) | Placebo at |
| | Total dose: 0 mg Spesolimab |

W: Week.

The multiple comparison procedure will then be implemented using optimal contrast tests, which control the family-wise type I error rate at a one-sided  $\alpha = 0.05$ . The optimal contrasts corresponding to each candidate model in the trial design stage are shown in <u>Table 7.4: 2</u>.

Table 7.4: 2 Contrast coefficients


| | Contrast coefficients for (total) dose | | | |
|---|---|---|---|---|
| Model | Placebo | Low dose: | Medium dose:<br>BI | High dose: |
| Linear | 0.592 | 0.254 | -0.085 | -0.761 |
| Exponential | 0.458 | 0.304 | 0.071 | -0.832 |
| Emax | 0.820 | -0.037 | -0.293 | -0.490 |
| SigEmax | 0.641 | 0.302 | -0.307 | -0.635 |
| BetaMod | 0.664 | 0.214 | -0.692 | -0.185 |

BI: Spesolimab total dose, i.e., sum of all loading and maintenance doses administered before week 8

For the final evaluation, these contrasts will be updated using the expected model means from the candidate set and the estimated variance-covariance matrix extracted from the MMRM model. The final contrasts will be presented in the CTR.

A non-flat dose response curve is established if at least one dose-response model is statistically significant, i.e., rejecting the null hypothesis of a flat dose-response curve

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

indicates a benefit of spesolimab over placebo. If a non-flat dose response is established, the statistically significant models from the above candidate set are refitted to the data without any parameter assumptions to generate new estimates for all model parameters.

The final model is derived as a weighted average over all significant model shapes. Here, the weights for each significant model  $(M_k)$  are given by

$$w(M_k) = \frac{\exp(0.5 \cdot \operatorname{AIC}(M_k))}{\sum_{i=1}^k \exp(0.5 \cdot \operatorname{AIC}(M_i))},$$

Where  $AIC(M_k)$  is the Akaike Information Criterion (AIC) of model  $M_k$ .

Estimates for each dose group will be calculated and final dose-response curve will be based on the final model. The confidence band for the final model will be based on parametric bootstrap approach by sampling from the multivariate normal distribution underlying the MMRM estimates and then fitting each of the models to each of these samples.

R code to perform the evaluations is available in Section 10.3.

The following displays are planned:

- Table of the updated contrast coefficients per dose group and candidate model, together with the MCPMod test statistics and p-values for each model and the critical value.
- For averaging model, figure of the dose-response curve and 95% confidence band for the bootstrap sampling.
- For all significant model shapes, figures of the dose-response curve plus 95% confidence band (of the predicated shape) and 95% CI per dose (estimated from MMRM).



c43421787-01



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.5 SECONDARY OBJECTIVE ANALYSIS

#### 7.5.1 Key secondary objective analysis

For part I, this section is not applicable as no key secondary endpoint has been specified in the protocol.

#### 7.5.2 Secondary objective analysis

For part 1, for each of the secondary endpoint, treatment policy will be used as the primary strategy to handle intercurrent events as for the primary endpoint.

### **Continuous secondary endpoints**

All secondary endpoints for part 1 are continuous endpoints, which will be analyzed using a MMRM approach based upon the model specification similar as described for the primary endpoint. Also, absolute change from baseline in IHS4 at week 8 is selected to use MCPMod to demonstrate a non-flat dose response curve.

SAS code for MMRM for the endpoint of IHS4:

The following SAS code will be used to calculate the MMRM.

**PROC MIXED** DATA=all at cl method=reml;

CLASS dt base categorical visit trt TNFi subject;

MODEL ept = TNFi dt base categorical visit\*trt base\*visit/ddfm=kr s CL;

REPEATED visit / subject= subject type=un r rcorr;

LSMEANS visit\*trt / pdiff=all om cl alpha=0.05 slice=visit;

RUN;




c43421787-01
c43421787-01



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### 7.7 EXTENT OF EXPOSURE

The exposure to study medication will be analyzed based on SAF. The number of subjects who received a dose of trial drug will be tabulated. The amount of total dose and duration of exposure will be summarized by descriptive statistics (N, mean, SD, minimum, median, maximum) for the overall on-treatment period, the loading stage, whole maintenance stage, maintenance stage I, maintenance stage II, maintenance stage III as described in <u>Table 6.1:1</u>. The duration of exposure will also be summarized with the following categories:

<= to <= 8 weeks</li>
> 8 weeks to <= 16 weeks</li>
> 16 weeks to <= to <= to <=</li>
to <=</li>

## 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the SAF following BI standards. Data will be summarized descriptively without any imputation based on data available.

As the onset time of an AE will not be collected in the trial, any AE which occurs on the same day as a treatment dose will be assigned to the on-treatment period defined in Table 6.1:1. For safety assessments by visits, if time is not collected, data on the same day of a treatment dose will be treated to be "prior treatment" except for scheduled local tolerability and post-dose vital signs assessments.

Off-treatment data will be listed only.

## 7.8.1 Adverse Events


Unless otherwise specified, the analyses of AEs will be descriptive in nature, which will include all on-treatment events up to week 8, week 16 treatment, as well as all events during the whole on-treatment period respectively. All analyses of AEs will be based on the number of subjects with AEs and NOT on the number of AEs.

AEs will be coded with the most recent version of MedDRA®. Patients will be analyzed according to the actual treatment received.

The analysis of AEs will be based on the concept of treatment emergent adverse events (TEAE). That means that all AEs occurring between first drug intake till 112 days after last drug intake will be assigned to the on-treatment period. All AEs occurring before first drug intake will be assigned to 'screening' and all AEs occurring after last drug intake + 112 days will be assigned to 'follow-up' (for listings only). For details on the treatment definition, see Table 6.1:1.

The exposure adjusted incidence rate (per 100 patient years) of a selected treatment emergent adverse event is defined as the number of patients experiencing the adverse event per

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

treatment group during time at risk divided by the total time of patients at risk in that treatment group to contribute the event to the analysis multiplied by 100 (per 100 patient years).

Time at risk [patient years] = (date of onset of AE– first treatment start date within that treatment period + 1) / 365.25

If, for a patient, the selected treatment emergent adverse event didn't occur during the above defined treatment period (per <u>Table 6.1:1</u>) then the time at risk will be censored at the earliest of date of death, last contact date per EoS page, or the end of the above defined treatment period.

For each selected treatment emergent AE, the exposure adjusted incidence rate will be calculated as:

Incidence rate [1/100 Patient years (pt-yrs)] = 100 \* number of patients with TEAE / Total TEAE-specific time at risk [patient years].

The analyses of AEs will be descriptive in nature. Analyses of AEs will be based on the exposure adjusted incidence rates (per 100 patient years), as well as the number of patients with AEs. System organ classes (SOCs) (if applicable) will be sorted according to the standard sort order specified by the European Medicines Agency (EMA), preferred terms (PTs) (if applicable) will be sorted by total frequency (within SOC).

For further details on summarization of AE data, please refer to "Handling and summarization of adverse event data for clinical trial reports and integrated summaries" (9.8) and "Handling of missing and incomplete AE dates" (9.1).

An overall summary of AEs will be presented. This overall summary will also include summary for the class of investigator reported AESIs.

The following are considered as AESIs (see Sec 5.2.6.1 of CTP):

- Systemic hypersensitivity including infusion reaction and anaphylactic reaction
- Severe infections (according to CTCAE grading in Section 15 of the ISF)
- Opportunistic and mycobacterium tuberculosis infections
- Potential Severe Drug Induced Liver Injury (DILI)
- Peripheral neuropathy


In addition, user defined adverse event concepts (UDAEC) identified through specific search criteria will be reported separately (see Table 7.8.1:1).

c43421787-01

Table 7.8.1: 1 Project MEDDRA search criteria for User Defined Adverse Events Concepts

| User-defined . | AE category | Category |
|---|---|---|
| Hypersensitivity | | |
| | Hypersensitivity ALL | All of the categories below |
| | Anaphylactic reaction, narrow | Narrow SMQ "Anaphylactic reaction" |
| | Angioedema, narrow | Narrow SMQ "Angioedema" |
| | Hypersensitivity, narrow | Narrow SMQ "Hypersensitivity" |
| Infections (serio | us/severe, opportunistic) | |
| | Infections 'ALL' | All of the categories below |
| | Opportunistic infections | Narrow SMQ "Opportunistic infections" |
| | Tuberculosis infections | Sub-BIcMQ "Tuberculosis related terms", narrow BIcMQ "Infections", narrow sub-search 8.2 "Tuberculosis related terms" |
| | Severe infections | SOC "Infections and infestations" with AETOXGR >= 3 OR AESEV = 'Severe'. Not derived for studies where both severity variables are collected. SOC "Infections and infestations" – AEs of at least |
| | Serious infections | severe CTCAE grade (>= 3) or any severe events SOC "Infections and infestations" with [AECOND: AESER =1] SOC "Infections and infestations" – SAEs |
| Malignancies | | |
| | Malignant tumours | Narrow sub-SMQ "Haematological malignant tumours", |
| | | Narrow sub-SMQ "Non-Haematological malignant tumours" |
| | | Narrow Sub-SMQ "Malignant tumours" |
| | Malignant skin tumours | Broad Sub-SMQ "Skin malignant tumours" |
| | Skin melanomas | HLT Skin melanomas (excl. Ocular) |
| | Non-melanoma skin cancer (NMSC) | Broad Sub-SMQ "Skin malignant tumours" excluding HLT Skin melanomas (excl. Ocular) |
| | Malignancies excluding non-<br>melanoma skin cancer<br>(NMSC) | Sub-SMQ "Malignant tumours" excluding NMSC defined above |
| 3 - point MACI | E for Monitoring | |
| | 3-point MACE for Monitoring | BIcMQ "Major Adverse Cardiovascular Events" wit<br>Narrow sub-search 1.1 "3-point MACE (part1/2) for<br>monitoring" |
| | | Narrow sub-search 1.2 "3-point MACE (part2/2) for monitoring" and AE outcome=fatal * |
| Depression | | |
| | Depression | Broad sub-SMQ "Depression (excl suicide and self-injury)" |
| Suicidal ideation | and behavior (SIB) | |
| | sub-SMQ "Suicide/self-injury" | sub-SMQ "Suicide/self-injury" |

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| User-defined AE category | | Category |
|---|---|---|
| DRESS# | | |
| | Narrow DRESS (Drug reaction with eosinophilia and systemic symptoms syndrome) | Narrow SMQ "Drug reaction with eosinophilia and systemic symptoms syndrome" |
| Peripheral N | europathy, Narrow | |
| - | Guillain-Barré Syndrome | Narrow SMQ "Guillain-Barré syndrome" |
| | Peripheral Neuropathy | Narrow SMQ "Peripheral Neuropathy" |
| | Demyelination | Narrow SMQ "Demyelination" |

<sup>\*</sup> This is achieved by retrieving all cases found either by running subsearch 1 in narrow scope (BIcMQ search ID 32019093) or subsearch 2 (BIcMQ serach ID 32019094).
# DRESS algorithmic search will be presented as a listing.

According to ICH E3 (9.9), in addition to Deaths and serious adverse events, 'other significant' AEs need to be listed in the clinical trial report. These will be any non-serious adverse event that led to an action taken with study drug (e.g. discontinuation or dose reduced or interrupted). An overall summary of adverse events will be presented.

The frequency of subjects with AEs will be summarized by treatment, primary system organ class and preferred term. AEs which were considered by the investigator to be drug related will be summarized separately. Separate tables will also be provided for subjects with SAEs, subjects with AEs leading to study drug discontinuation, subjects with AESIs, subjects with other significant AEs (derived based upon ICH E3 (9.9)), User-defined Adverse Event Concepts (UDAEC) (Table 7.8.1:1) and serious UDAEC. AEs will also be summarized by maximum intensity based on the CTCAE grading system.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5% (in preferred terms) will be summarized by treatment, primary system organ class and preferred term. The frequency of subjects with SAEs will also be summarized.

## 7.8.2 Laboratory data


The analyses of laboratory data will be descriptive in nature and will be based on BI standards (9.3). The up to Week 16 and overall on-treatment period for laboratory analyses will be provided. Note that data from the central laboratory will be used for all displays described below, unless otherwise specified.

For continuous safety laboratory parameters, normalized values will be derived.

Normalization means transformation to a standard unit and to a standard reference range. The process of normalization, handling of repeat values at the same visit for by-visit displays, as well as standard analyses for safety laboratory data are described in the BI guidance for the Display and Analysis of Laboratory Data. All analyses considering multiple times of the ULN (as described below) will be based on standardized and not normalized values. For continuous


c43421787-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

safety laboratory parameters, differences to baseline will be calculated. For all outputs, the last assessment before the first treatment at Day 1 is chosen as the baseline value.

Only patients with at least one available post-baseline value will be included in the analysis of an individual laboratory parameter. All individual laboratory data will be listed. Values outside the reference range will be flagged.

For derivation of the last value, the minimum value, and the maximum value, all values during the on-treatment period will be considered. These will be derived for analysis of laboratory, vital signs and local tolerability data. For identification of potentially clinically significant abnormal laboratory values, all values during on-treatment period will also be considered.

Descriptive statistics of laboratory values over time and for the difference from baseline ontreatment will be based upon normalized values, including summaries of the last value on treatment, the minimum value on treatment and the maximum value on treatment and corresponding change from baseline. Graphical displays via box plots/line plots will be produced for the last value, minimum and maximum value on treatment for each continuous laboratory endpoint.

Laboratory values will be compared to their reference ranges; shift tables will be provided for the number of patients with a specific CTCAE grade at baseline versus the CTCAE grade at the last measurement on treatment, as well as the worst grade on treatment; laboratory parameters with exception to this display type are described in the company standards (9.10). These analyses will be based on converted laboratory values. The display of laboratory data using the CTCAE grades will be done based on BI standards (9.10).

Potentially clinically significant abnormalities will be identified based on BI standard rules which are based on converted lab values, i.e. using SI units. These rules will be listed in the SDL appendix of the CTR. Frequency tables will summarize the number of patients with potentially clinically significant abnormalities. Patients having an abnormal lab value at baseline will be presented separately. A separate listing will present potentially clinically significant abnormal lab values; for each functional lab group all patient's lab values will be listed, if there exists at least one lab value with clinically significant abnormality within the group.

The frequency of patients with AST or ALT elevations  $\geq 3xULN$ ,  $\geq 5xULN$ ,  $\geq 10xULN$ , and  $\geq 20xULN$  will be displayed based on standardized laboratory values. To support analyses of liver related adverse drug effects, the frequency of subjects with AST and/or ALT  $\geq 3xULN$  combined with the elevation of total bilirubin  $\geq 2xULN$ , from samples drawn within 30 days of each other, will be displayed, stratified by alkaline phosphatase < 2xULN and  $\geq 2xULN$  (a subject can potentially be in both alkaline phosphatase strata in case of multiple AST/ALT and bilirubin elevations). The start of the 30-day time span is triggered by each liver enzyme elevation above the defined thresholds. This analysis will be based on standardized laboratory values.


Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

A graphical analysis of ALT and total bilirubin will be performed: the so-called eDISH plot. The peak total bilirubin is presented as a fold increase over the ULN against the peak ALT as a fold increase over the ULN, on a log10 scale. The measurements displayed for total bilirubin and ALT may, or may not, occur on the same date. Two reference lines, 2xULN for total bilirubin and 3xULN for ALT, are drawn onto the graph to divide the plane into four quadrants. Normal cases are in the lower left quadrant, potential DILI cases are in the upper right quadrant (potential Hy's Law quadrant), while the lower right quadrant is known as the Temple's corollary range (ALT  $\geq 3xULN$  and total bilirubin < 2xULN). The display will be repeated for AST and total bilirubin.

The frequency of subjects with AST and/or ALT  $\geq$  3xULN combined with the elevation of INR  $\geq$  1.5xULN, from samples drawn within 30 days of each other, will be displayed. The start of the 30-day time span is triggered by each liver enzyme elevation above the defined thresholds. This analysis will be based on standardized laboratory values.

A graphical analysis of ALT and INR will be performed. The peak INR is presented as a fold increase over the ULN against the peak ALT as a fold increase over the ULN, on a log10 scale. The measurements displayed for INR and ALT may, or may not, occur on the same date. Two reference lines, 1.5xULN for INR and 3xULN for ALT, are drawn onto the graph to divide the plane into four quadrants for better visual representation; normal cases are in the lower left quadrant. The display will be repeated for AST and INR.

An additional display will be produced for the frequency of patients with an elevation of the ALT and/or AST  $\geq$  3-fold ULN, and with the appearance of one or more of the following TEAE:

• Fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

An occurrence is flagged if, within  $\pm$  7 days of the onset of an AST and/or ALT elevation  $\geq$  3-fold ULN (including events which start or are ongoing through this interval [i.e., including also assessment on the AE stop in addition to the start date]), at least one of the following TEAE terms (excluding PT terms on the secondary path) is observed:

- ADAE.AEHLT = "Gastrointestinal and abdominal pains (excl oral and throat)";
- ADAE.AEDECOD in ("Vomiting", "Fatigue", "Nausea", "Pyrexia", "Right upper quadrant pain", "Abdominal pain upper", "Upper abdominal tenderness");
- ADAE.CQ16NAM = "Skin Rash (BIcMQ narrow);


An occurrence is also flagged if a >5% proportion in the ratio of eosinophils to total white blood cells is observed in the same sample as the detected AST/ALT elevation.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analyzed as such.

# 7.8.3 Vital signs

Descriptive statistics and graphical display are planned for this section of the report.

The analyses of vital signs (blood pressure, pulse rate, body temperature, respiratory rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided, including the last value, the minimum value and the maximum value during on-treatment period.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analyzed as such.

#### 7.8.4 ECG

Abnormal findings in 12-lead ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analyzed as such.

## 7.8.5 Local Tolerability

Local tolerability will be summarized during on-treatment period and by visit, with the frequency and percentage of patients who experienced any symptoms by severity/intensity.

## 7.8.6 Acne Episodes


In the final analysis, the occurrence and characteristics of historical acne episodes will be summarised by treatment with frequency and percentage of patients. The characteristics of any acne episodes which occur during the treatment period will be displayed overall; separate displays of the characteristics of those acne episodes which had a) a suspected medical history risk factor, b) a suspected concomitant medication risk factor, and c) a relatedness to spesolimab, will also be presented. If only few records for the acne episodes, listings will be provided instead of summary tables.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### 7.9 OTHER ANALYSIS

# 7.9.1 Biomarker analyses

The following biomarkers will be analysed and reported as a part of the CTR:

•

For the analysis of values below the lower limit of quantification (LLOQ) or above the upper limit of quantification (ULOQ) will be handled as follows:

Values < LLOQ and values > ULOQ that are reported as numerical values, will be kept as such. Entries reported as text (i.e. "< LLOQ" or "> ULOQ") and for which no value is provided, will be replaced by:

For < LLOQ: 0.5\*LLOQ</li>For > ULOQ: ULOQ.

Results on other biomarkers (e.g.

of the

data. In case they are reported outside the CTR the analysis will be defined in a separate document (otherwise the analysis will be described in the CTR).

For the analysis of biomarkers, log transformed data will be used where deemed necessary.

# 7.9.2 PK/PD analyses


No PK parameters will be calculated.

The descriptive analysis of Spesolimab plasma concentrations will be based on the SAF.

# **Exclusion of PK concentrations**

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times.

Further details are given in (9.7). No formal analysis of pharmacokinetic/pharmacodynamic relationships is planned.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Any further exploratory analyses, if done, will be described in the CTR or in a separate report.

# 7.9.3 Immunogenicity


The ADA status and titer as well as frequency of patients with ADA to Spesolimab will be presented by visit. Descriptive statistics of ADA titer (for ADA positive patients, when available) will be provided by visit. The number of subjects with ADA status positive/negative at any time will also be presented. ADA parameters (e.g. treatment-induced ADA positive subjects, transient ADA response and persistent ADA response) will also be presented by visit and cumulatively for the overall study duration. Further exploratory assessments of the ADA data will be performed once data is available and these will be described, if done, in the CTR.

Further analyses based on ADA data may be performed such as

- efficacy-based subgroup analysis for selected subgroups in <u>Table 6.5: 1</u> for the following groups
  - ADA positive and ADA negative subjects (at Week 8 and Week 16 visit), or
  - NAb positive and NAb negative subjects (at Week 8 and Week 16 visit)
- Safety-based subgroup analysis (using e.g. hypersensitivity safety events) for the following groups
  - ADA positive and ADA negative subjects (at any time), or
  - NAb positive and NAb negative subjects (at any time), or

before ADA development (including subjects with events either before their first ADA positive sample or without ADA positive sample throughout) and after ADA development (including subjects with events from the time point of their first ADA positive sample onwards). This approach takes into account the time when ADA actually developed and when the safety event occurred in relationship to ADA.

c43421787-01

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be released for interim analysis according to the details specified in the logistics plan.

Once the last patient has completed their *End-of-Treatment (EOT) visit* and all corresponding data has been entered and cleaned to the level documented in the "Data Delivery Request" (DDR) form, the data will be declared ready to be unblinded via the "Data Ready to be Unblinded and/or Final Trial Closure Notification" (RUN) form. Then the treatment information will be released for analysis.

The data collection for the off-treatment residual effect period until the End-of-Study (EoS) / Follow-Up visit will continue into the unblinded trial database. Once trial data collection has been completed and all data has been entered and cleaned as documented on the RUN form, a final data lock will be performed.

After the release of treatment information, it is expected that only trial data related to the off-treatment residual effect period will be entered and changed. Therefore, after the timepoint of release of treatment information, all changes affecting trial data up to the End-of-Treatment (EoT) visit will be documented and summarized in the CTR.

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 9. REFERENCES


| 9.1 | <i>BI-KMED-BDS-HTG-0035</i> : "How to Guide: Handling of Missing and Incomplete AE dates", current version, KMED. |
|---|---|
| 9.2 | BI-KMED-TMCP-HTG-0025: "How to Guide: Standards and Processes for Analyses Performed within Clinical Pharmacokinetics/Pharmacodynamics", current version, KMED. |
| 9.3 | BI-KMED-BDS-HTG-0042: "How to Guide: Handling, Display and Analysis of Laboratory Data", current version, KMED. |
| 9.4 | <i>Pinheiro J, Bornkamp B, Bretz F.</i> Design and analysis of dose-finding studies combining multiple comparisons and modelling procedures. J Biopharm Stat 16 (5), 639-656 (2006). |
| 9.5 | <i>Pinheiro J, Bornkamp B, Glimm E, Bretz F.</i> Model-based dose finding under model uncertainty using general parametric models. Stat Med 33 (10), 1646 – 1661 (2014). |
| 9.6 | BI-VQD-12045_40-413: "Identify and Manage Important Protocol Deviations (iPD) ", current version, group / owning department "Med Clinical Development & Operations", DMS for controlled documents. |
| 9.7 | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON. |
| 9.8 | 001-MCG-156: "Handling and summarisation of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON |
| 9.9 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version, EMA webpage. |
| 9.10 | <i>BI-KMED-BDS-HTG-0036</i> : "How to Guide: CTCAE Grading for Laboratory Values", current version, KMED. |
| 9.11 | Heinze G, Schemper M. A solution to the problem of separation in logistic regression. Statistics in Medicine 21: 2409-2419 (2002). |
| 9.12 | Firth D. Bias reduction of maximum likelihood estimates. Biometrika 80, 27–38 (1993) |
| 9.13 | Greenland S, Robins M. Estimation of a common effect parameter from sparse follow-up data, Biometrics 41, 55-68, 1985 |
| 9.14 | Sato T. On the Variance Estimator of the Mantel-Haenszel Risk Difference, Biometrics, 45, 1323–1324, 1989, letter to the editor. |

c43421787-01

| 9.15 | Zouboulis C.C., Tzellos T., Kyrgidis A., Jemec G.B.E., Becha |
|---|---|
| | F.G., et al. European Hidradenitis Suppurativa Foundation |
| | Investigator Group. Development and validation of the |
| | International Hidradenitis Suppurativa Severity Score System |
| | (IHS 4), a novel dynamic scoring system to assess HS severity. Br |
| | J Dermatol. 2017 Nov; 177 (5): 1401-1409. |
| 9.16 | Rubin, DB. Multiple Imputation for Nonresponse in Surveys. New |
| | York: John Wiley &Sons. 1987. [R12-2378] |

c43421787-01



c43421787-01

c43421787-01



c43421787-01



c43421787-01



c43421787-01



c43421787-01

| Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. |
|---|

c43421787-01





c43421787-01



c43421787-01



c43421787-01



Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 11. HISTORY TABLE

Table 11: 1 History table


| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1.0 | 13-08-2024 | | None | This is the final TSAP. |